CLINICAL TRIAL: NCT00347022
Title: A Clinical Study of Xenetix 300 in Multislice Computed Tomography (CT) Pediatric Indications
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Guerbet (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: ISO-44-008
Record Dates: First submitted 2006-06-30; First posted 2006-07-04 (Estimated); Results first posted 2013-04-09 (Estimated); Last update posted 2013-04-09 (Estimated); Status verified 2013-04

CONDITIONS: Diagnostic Imaging
Keywords: Multislice computed tomography (MSCT)indications
MeSH Terms: interventions — iobitridol; iodixanol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- Xenetix (Experimental): The patient receive one injection of Xenetix 300 (300 mg of iodine/ml)
  Interventions: Drug: Xenetix
- Visipaque (Active Comparator): The patient receive one injection of Visipaque 270 (270 mg of iodine/ml)
  Interventions: Drug: Visipaque

INTERVENTIONS:
Drug: Xenetix — 300 mg of iodine/ml
  Arms: Xenetix
Drug: Visipaque — 270 mg of iodine/ml
  Arms: Visipaque

SUMMARY:
This is a clinical study of Xenetix 300 in Multislice Computed Tomography (MSCT) in pediatric indications.

ELIGIBILITY:
Inclusion Criteria:

* Child aged 1 year or above and 16 years or under
* Patients with normal renal function (creatinine clearance > 60 ml/min/1.73 m2)
* Patient requiring MSCT with contrast medium injection for diagnosis
* Patient who has a blood sample planned in the 24 hours preceding the MSCT scan
* Female patient with childbearing potential must have effective contraception (contraceptive pill or intrauterine device), be surgically sterilized or blood beta human chorionic gonadotropin (ßHCG) will be tested prior to product injection.
* Parent(s) of the patient (and child with sufficient intellectual maturity) provided his/her/their written informed consent for their child to participate in the trial.
* Patient with national health insurance

Exclusion Criteria:

* Patients who have received diuretic or biguanide treatment during the 48 hours preceding the MSCT scan.
* Patient with known allergy to iodinated contrast agent.
* Patient treated with nephrotoxic drugs within one week before first blood sample
* Patients planned to either undergo surgery or receive chemotherapy within 72 hours post injection (ie: before the blood test 72 hours post injection)
* Patient received or planned to receive an iodinated contrast agent during 48 hours preceding the MSCT scan.
* Breast feeding patient.
* Pregnant patient.
* Patient already included in this trial
* Patient included in another clinical trial involving an investigational drug.
* Patients whose degree of cooperation is incompatible with carrying out the study

Ages: 1 Year to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 145 (Actual)
Dates: Start 2006-05; Primary Completion 2009-04 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Corinne Dubourdieu, PhD, Study Chair — Guerbet
Locations (1):
- CHU Charles Nicolle, Rouen, France

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First patient first visit = 30/05/2006 Last patient last visit = 14/04/2009 Location = radiological department (Hospitals)
Pre-assignment Details: Any patient having a creatinine clearance < 60ml/min/1.73m² at time of baseline blood sample and/or positive beta HCG (Human Chorionic Gonadotropin) within 48h before contrast medium administration was considered as immediate withdrawal from trial
Groups:
- Xenetix: Patient will receive one injection of Xenetix 300
- Visipaque: Patient will receive one injection of Visipaque 270
Period: Overall Study
Arm/Group | Xenetix | Visipaque
Started | 74 | 71
Completed | 62 | 66
Not Completed | 12 | 5

BASELINE CHARACTERISTICS:
Groups:
- Xenetix: Patient will be injected with Xenetix 300
- Visipaque: Patient will be injected with Visipaque 270
- Total: Total of all reporting groups
Arm/Group | Xenetix | Visipaque | Total
Number analyzed (Participants) | 74 | 71 | 145
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 74 | 71 | 145
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 8.7 (4.8) | 8.1 (4.7) | 8.4 (4.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 28 | 59
  Male | 43 | 43 | 86
Region of Enrollment [Number; unit: participants]
  France | 59 | 56 | 115
  Austria | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Creatinine Clearance
Description: The variation of creatinine clearance before and after the product injection was measured
Time Frame: between 48h before the contrast medium administration and 72h +/-12h after contrast medium administration
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Xenetix | Visipaque
Number analyzed (Participants) | 62 | 66
percent change | 1.1 (19.7) | 1.9 (22.0)

ADVERSE EVENTS:
Groups:
- Vispaque: Patient will be injected with Visipaque 270
Arm/Group | Xenetix | Vispaque
Serious Adverse Events (participants affected / at risk) | 5/74 | 4/71
Other Adverse Events (participants affected / at risk) | 11/74 | 13/71
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Xenetix (N=74) | Vispaque (N=71)
Surgery of vesical wound (Surgical and medical procedures) | 0 (0) | 1 (1)
Myelofibrosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Meningitis (Nervous system disorders) | 0 (0) | 1 (1)
Ent surgery (Surgical and medical procedures) | 0 (0) | 1 (1)
Mastoidectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Operation of the mediastinal haematoma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Abdominal operation (Surgical and medical procedures) | 1 (1) | 0 (0)
Inflammatory syndrome (General disorders) | 1 (1) | 0 (0)
Pyramidal syndrom (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Xenetix (N=74) | Vispaque (N=71)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Increase of creatinine (Investigations) | 4 (4) | 7 (7)
Allergic cutaneous reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Cutaneous eruption (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Leukoencephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fever (General disorders) | 1 (1) | 2 (2)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Extravasation (General disorders) | 1 (1) | 0 (0)
Oedema neck and face (General disorders) | 1 (1) | 0 (0)
Tracheitis (Infections and infestations) | 1 (1) | 0 (0)
Vagal discomfort (Nervous system disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Warmth at the site of injection (General disorders) | 0 (0) | 1 (1)
Red papules on the arm (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
* Draft of publication to be submitted by the coordinating investigator (no more than 6 months after getting study results) to sponsor and other investigators for review at least 1 month before the submission to the scientific review. Comments to be reviewed and approved by the coordinating investigator and sponsor.
* Each investigator agrees not to publish the comparison of the renal tolerance involving only the patients he/she has included.